CLINICAL TRIAL: NCT02719509
Title: Prospective Evaluation of the Utility of Bedside Cardiac Ultrasound for Undifferentiated Chest Pain and Shortness of Breath in the Emergency Department
Brief Title: Emergency Department Cardiac Ultrasound
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HSR # 15-4092
Record Dates: First submitted 2016-02-04; First posted 2016-03-25 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Chest Pain; Dyspnea
MeSH Terms: conditions — Chest Pain; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational Cohort: All emergency department patients who had a cardiac ultrasound performed as part of their diagnostic workup
  Interventions: Procedure: Cardiac Ultrasound

INTERVENTIONS:
Procedure: Cardiac Ultrasound

SUMMARY:
This is a prospective observational study evaluating the diagnostic utility of cardiac ultrasound in patients who present to the emergency department with undifferentiated chest pain or shortness of breath. Emergency department providers will be interviewed before and after the completion of a cardiac ultrasound to determine if the ultrasound resulted in any changes in management. Other outcomes include determination of incidence of unexpected findings.

DETAILED DESCRIPTION:
Bedside cardiac ultrasound is performed regularly in the emergency department to assess patients who present with undifferentiated chest pain or shortness of breath. Utility of cardiac ultrasound in this setting is emerging as standard of care. Cardiac ultrasound can rapidly provide essential information about the presence or absence of multiple cardiopulmonary pathologies. Cardiac ultrasound is safe, immediately accessible, and gives providers data regarding their patients in real-time.

While cardiac ultrasound is common practice in emergency departments, the diagnostic utility of this test has been difficult to study. There are few studies in the literature that describe its utility in evaluating specific diagnoses. These studies have evaluated the use of cardiac ultrasound in diagnosing acute cardiogenic pulmonary edema, aortic dilation/aneurysm, acute coronary syndrome, and acute heart failure.

The purpose of this study is to evaluate the utility of cardiac ultrasound in patients who present to the emergency department with undifferentiated chest pain or shortness of breath. This study will evaluate several parameters including how the cardiac ultrasound contributes to provider's management plan and assessment of the patient's diagnosis.

This is a prospective observational study design. The investigators will prospectively enroll eligible consecutive patients who present to the emergency department with undifferentiated chest pain or shortness of breath. Patients will be included if a provider has ordered (or is planning on ordering) a cardiac ultrasound as part of the patient's diagnostic workup. Research associates will screen for these two chief complaints and will then approach the ED provider and ask if they ordered or are planning to order a cardiac ultrasound. ED providers may also contact research associates to enroll patients that meet the study criteria.

Pre-ultrasound assessment: After eligibility is determined, a research associate will approach the provider directly involved in the patient's care (Resident or Staff). The provider completing the data collection forms does not need to be the provider who ordered or performed the ultrasound. The provider completing the forms will be an Emergency Medicine 2nd year level resident or above. The provider filling out the data collection form will fill out the pre-ultrasound assessment prior to reviewing the cardiac ultrasound images (either in real-time or on the computer after the ultrasound is completed). The provider will fill out a data collection form that asks about the most likely diagnosis, expected ultrasound findings, and current management plan.

After the ultrasound is completed the same provider will be asked about the most likely diagnosis, observed ultrasound findings, and any new management changes.

Other clinical data that will be collected will include demographic data, vital signs, relevant co-morbidities, imaging results, and lab results from the emergency department visit.

ELIGIBILITY:
Inclusion Criteria:

* ED patients with a chief complaint of chest pain or shortness of breath
* Cardiac Ultrasound ordered by provider as part of diagnostic workup

Exclusion Criteria:

* All providers have already reviewed the ultrasound images (unable to obtained pre- ultrasound assessment)
* Age < 18
* Known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with undifferentiated chest pain or shortness of breath who have a cardiac ultrasound ordered by the emergency provider as part of the diagnostic workup
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of management changes | 6 hours
  Approximate duration of the emergency department visit

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Klein, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided